CLINICAL TRIAL: NCT00243685
Title: Application of the Microculture Kinetic (MiCK) Assay for Apoptosis to Drug Testing Sensitivity of Solid Tumors
Brief Title: Chemotherapy Drug Sensitivity Microculture (MiCK) Assay for Apoptosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pierian Biosciences (Industry)
Responsible Party: Cary Presant, MD, DiaTech Oncology
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 20050113
Record Dates: First submitted 2005-10-20; First posted 2005-10-24 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Breast Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Sarcoma, Soft Tissue
Keywords: Chemosensitivity; Chemotherapy; Lung cancer; Ovarian Cancer; Breast Cancer; Sarcoma; Apoptosis; MiCK Assay; New Technology; Patients with pathological diagnoses of breast, lung, and ovarian adenocarcinomas and soft tissue sarcoma
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Sarcoma | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- II and III (Experimental)
  Interventions: Other: Laboratory Assay; Other: Mick Assay

INTERVENTIONS:
Other: Laboratory Assay — Chemotherapy
  Other Names: Comparison of differnt drugs
Other: Mick Assay — Chemotherapy doctor determined from results
  Other Names: Chemotherapy

SUMMARY:
DiaTech is a private company performing patient specific cancer chemosensitivity testing for patients and physicians. DiaTech Oncology is doing this clinical study to see if an experimental new technology called the microculture kinetic (MiCK) assay will predict treatment outcome and can help to direct the chemotherapy of cancer subjects. This study is focused on subjects diagnosed with breast, ovarian, lung, and colon malignancies and low-grade lymphomas.

Study Objectives:

* To evaluate the ability of the MiCK assay to predict the outcome of chemotherapy of cancer patients.
* To evaluate the ability of the MiCK assay to guide chemotherapy of cancer patients.

DETAILED DESCRIPTION:
Application of the Microculture Kinetic (MiCK) Assay for Apoptosis to Testing Drug Sensitivity of Solid Tumors DiaTech Oncology, LLC

----------------------------------------------------------- 1.0 Background and Rationale: Despite the use of aggressive treatment protocols, less than 10% of cancer patients with an advanced disease respond to the therapy. There is a variety of different cancer drug regimens, all of which have approximately the same probability of clinical effectiveness. Identification of those patients who will or will not respond to a specific chemotherapy is important for making decisions regarding chemotherapy regimens as well as alternative management approaches. A laboratory test that could help to determine the sensitivity of an individual patient's tumor cells to specific chemotherapeutic agents would be valuable in choosing the optimal chemotherapy regimen for that patient with an expectation of increasing the response rate to the therapy. Several types of in vitro assays that measure tumor cell survival following exposure to cytotoxic agents have been evaluated for their ability to predict chemotherapy outcomes. As a group, these assays are referred to as drug resistance assays. In a resistance assay, the surviving tumor cells can be detected directly by their exclusion or metabolism of specific dyes. Alternatively, since some of tumor cells are proliferating, their survival can be detected by measurement of DNA synthesis by radiolabeled precursor incorporation or demonstration of clonogenic potential by growth into colonies in semi-solid culture medium. In several clinical studies, these assays were useful in detecting drug resistance and in predicting a poor prognosis for cancer patients. However, these resistance assays cannot detect sensitivity of an individual patient's tumor cells to a specific drug. Therefore, new methods determining drug-sensitivity of the tumor cells of an individual patient and, thus, capable of both predicting a positive treatment outcome and guiding chemotherapy, would be of significant value.

Recently, Dr. Kravtsov has developed an automated microculture kinetic (MiCK) assay for measuring drug induced apoptosis in tumor cells1-4. Apoptosis is a distinct mode of cell death which occurs under physiological conditions and yet can be induced in malignant cells by chemical and physical factors including antitumor drugs5-7. During the last decade, it has been recognized that chemotherapeutic agents exert their antitumor activity by triggering apoptosis in susceptible tumor cells8-17. This implies that the MiCK assay for apoptosis provides a mechanism-based approach to studying effects of cytotoxic agents on tumor cells. Unlike "resistance" assays that measure a fraction of cells surviving drug exposure, the MiCK assay measures a fraction of tumor cells killed by a chemotherapeutic agent via mechanism of apoptosis. Therefore the MiCK assay determines drug sensitivity, rather than resistance. Recently the MiCK assay has been shown to predict complete remission rate and survival in acute myeloid leukemia patients better than clinical criteria did18-20. In a limited study, the MiCK assay has been used to direct chemotherapy of the leukemia patients 21.

The MiCK assay has also been used to study drug-induced apoptosis in solid tumors, including neuroblastoma and colon adenocarcinoma cell lines22-23. More recent data accumulated by DiaTech has demonstrated that the MiCK assay can detect drug induced apoptosis in primary cultures of tumor cells isolated from patients with ovarian carcinoma, gastric carcinoma, metastatic breast cancer and high grade soft tissue sarcoma. Based on these data, we suggest that the MiCK assay may be used to detect drug sensitivity profiles of individual patients with various types of solid tumors. This, in turn, may provide a way to tailor chemotherapy to an individual patient's drug sensitivity profile, and, thus, improve treatment outcomes, decrease adverse effects of the chemotherapy, increase the quality of patient's life, and reduce the treatment cost.

2.0 Study Objectives: 2.1 To evaluate the ability of the MiCK assay to predict the outcome of chemotherapy of cancer patients.

2.2 To evaluate the ability of the MiCK assay to guide chemotherapy of cancer patients.

3.0 Patient Population:

3.1 Inclusion criteria: 3.1.1 Patients with pathological diagnoses of breast, lung, and ovarian adenocarcinomas and soft tissue sarcoma.

3.1.2 Patients with de novo malignancies and no previous chemotherapy 3.1.3 Patients with advanced refractory malignancies who received no more than 2 standard chemotherapy treatment protocols.

3.1.4 Patients of any age group. 3.1.5 Patients must have tumor which is accessible and agree to undergo biopsies, or drainage of effusions.

3.1.6 Patients for whom chemotherapy is a treatment option. 3.2 Explanations: We anticipate that newly diagnosed patients will be mostly used to evaluate the ability of the MiCK assay to predict the outcome of the chemotherapy (Objective #2.1) and to establish criteria correlating numerical response in the MiCK assay with probability of the clinically established complete remission. The patients with refractory malignancies will be mostly used to evaluate the ability of the MiCK assay to guide cancer chemotherapy (Objective #2.2). Patients will be seen and managed as outpatients or inpatients, depending on a clinical standard of the institution.

3.3 Exclusion criteria: 3.3.1 Patients with symptomatic/uncontrolled parenchymal brain metastasis and not accessible tumors.

3.3.2 Patients with meningeal metastasis. 3.3.3 Patients for whom chemotherapy clinically is not indicated. 3.3.4 Pregnancy. During the course of the study, all patients of childbearing potential should be instructed to contact the treating physician if they suspect they might have conceived a child; for females, a missing or late menstrual period should be reported to the treating physician. If pregnancy is confirmed by a pregnancy test, the patient must not receive study medication and must not be enrolled into the study or, if already enrolled, must be withdrawn from the study. If a male patient is suspected of having fathered a child while on the study drugs, the pregnant female partner must be notified and counseled regarding the risk to the fetus. Pregnancy during the course of this study will be reported to the Principal Investigator as a serious adverse event. Women of child bearing potential are defined to include any female who has experienced menarche and has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not post-menopausal (defined as amenorrhea for more than 12 consecutive months); these includes also females using oral, implanted, or injectable contraceptive hormones, mechanical devices, or barrier methods to prevent pregnancy.

4.0 Treatment Plan: 4.1 For the patients involved under the Study Objective (2.1), treatment protocol for an individual will not be influenced by the results of the MiCK assay for that patient. Oncologists will be blinded of the results of the MiCK assay and the patients will be treated according to a standard treatment protocol. When available, actual clinical response to the treatment will be compared with that predicted by the MiCK assay.

4.2 For the patients involved under the Study Objective (2.2), treatment protocol for an individual patient will be designed based on the results of the MiCK assay for that patient. The drug with the best activity in the assay will be used to treat the individual patients. If more than one drug is equally active, the patient will receive the active drug in a class he/she has not received before. If no drug is found to have activity (insensitivity in the assay), the patients will be treated on an empiric basis with a class of drug he/she never received in the past.

5.0 Definition of Clinical Response 5.1 All patients will be evaluated for clinical response to chemotherapy as per standard protocol established for a specific malignancy.

5.1.1 Complete Remission is defined as total disappearance of clinically and radio logically detectable disease for at least four weeks.

5.1.2 Partial Response is defined as at least 50% reduction of all measurable tumor lesions as measured by the sum of products of the perpendicular diameters of the greatest dimensions of measurable lesions, with no new lesions appearing for at least four weeks.

5.1.3 Stable Disease is defined as a reduction by less than 50% or increase by less than 25% in the size of the tumor lesions, with no new lesions appearing.

5.1.4 Progressive Disease is defined as appearance of any new tumor lesions or increase of 25% or more in the sum of products of the perpendicular diameters of the greatest dimensions of measurable existing lesions.

6.0 Definition of the drug response in the MiCK assay. 6.1 In the MiCK assay, the extent of drug-induced apoptosis is measured in Kinetic Units (KU) on a scale from 0 to 16 (Blood, 1998). Apoptotic responses in KU will be calculated for each dose of a tested drug or drug combination. The maximal numerical response induced by a drug will be considered the "best apoptotic response" to the drug.

6.1.1 Under the Study Objective (2.1), the "best apoptotic response" to the drug will be compared to the clinical response to the drug to establish a numerical value of the in vitro response discriminating drug-sensitive and drug-insensitive tumors (establishing a numerical cut-off of sensitivity). From our experience with establishing cut-off values of drug sensitivity for acute leukemia, 25-30 patients should provide a sufficient statistical power for getting a significant discriminator. These 25-30 patients will be fed from both patients participating under Study Objective (2.1) and Study Objective (2.2). After the numerical cut-off for sensitivity is established, it will be applied to a cohort of patients who received treatment with the drug to compare responses predicted in the MiCK assay to the actual clinical responses. This second part of the study will have two legs: (a) "prospective" (using 30-35 patients entering the study after establishing the discriminator, and (b) "retrospective" (using an available database of the patients who received treatment in the past and who's clinical response to the chemotherapy is known).

6.1.2 For the patients participating under the Study Objective (2.2), a drug inducing the highest "best apoptotic response" will be considered the best active drug and will be recommended for including in the treatment protocol. Only drugs with the numerical value of the "best apoptotic response" exceeding a certain threshold should be expected to induce a complete remission. In the beginning of the study, such a threshold will be judged based on the results of the previous leukemia study19-22. As first 25-30 patients enter the study, the thresholds will be established for solid tumor patients as described in (6.1.1) and used thereafter. Considering that these 25-30 patients will be fed from both patients participating under Study Objective (2.1) and Study Objective (2.2), we expect to have first statistical correlations available no later than 3-4 months after the study begins.

6.1.3 Drug selection for testing against tumor cells will be based on the previous chemotherapy history of an individual patient with consideration of the future treatment plans. The drugs will be selected from a compendium of agents recommended for the treatment of the patient's malignancy.

7.0 Statistics 7.1 We estimate that sufficient statistical power will be obtained with approximately 50-60 patients with successful MiCK assays. A successful MiCK assay is defined as an assay for which a sufficient number of viable tumor cells could be isolated from the submitted pathologic material. For correlations between the patient's sensitivity profiling in the MiCK assay and clinical responses, the patients will be evaluated as the whole group as well as stratified based on the type of malignancy. The latter will depend on the number of patients with specific tumor types available for the study.

7.2 In order to discriminate between the drug-sensitive and drug insensitive tumor cell populations, the best responses to each agent will be compared in a receiver operator characteristic (ROC) analysis as well as logistic regression analysis with attainment of CR (CR vs No CR). Based on the best combination of statistical sensitivity, specificity, and p value, thresholds demarcating drug sensitivity and insensitivity will be established. The Fisher's exact test, chi-square test and analysis of variance method will be employed to test the correlation between the clinical response results and other clinical variables. For lifetime data analyses, Kaplan-Meier estimates of survival will be used. Other statistical techniques may also be implied if found useful.

8.0 Specimen collection, purification of tumor cells and sensitivity testing 8.1 Specimen collection must be performed as per related DiaTech Standard Operating Procedures (SOP).

8.1.1 Collection of a Solid Tumor Biopsy Specimen is performed under sterile conditions, using excision biopsy technique, to obtain at least 2 cm3 of viable tumor tissue. The more viable tumor tissue is submitted for the study, the more chemotherapeutic agents can be tested against the tumor cells. Effusion specimen (peritoneal fluid, pleural fluid and effusions from other anatomical sites) should be collected in a commercial sterile container/bag with added Sodium Heparin (10 U/ml) to prevent clotting. The sample size should not be less than 500 ml. The specimen should not be fixed, or frozen.

8.1.2 Transportation: seal the transport tube/container/bag tightly. Label specimen with institution, patient name, date and time of collection, and anatomical site of collection. Place the transport tube/container/bag on ice pack (blue ice). Ice pack must be frozen before placing it to the container. Fill out the Study Requisition form and include with the transportation container.

8.1.3 Place the 50 mL tubes or a container inside the zip-lock bag and seal. Place specimen and Cold Pak (blue ice) in a transport box. Place completed patient information forms and specimen transport box into FedEx plastic "Diagnostic Specimen Envelope" and seal. Complete and affix the FedEx Airbill to the outside of the Diagnostic Specimen Envelope. Be sure that the airbill is marked "FedEx Priority Overnight" delivery. Put $5 value on the FedEx Airbill. Indicate "Human tissue for diagnostic studies" in the appropriate section of the FedEx Airbill. Call DiaTech Oncology at (514)-398-5174 (Steve Moisan, lab manager) or (514)-398-5154 (general lab) with the Fed Ex Tracking Number. DiaTech must receive the specimen within 24 hours of collection. Specimens sent on Friday must be marked for Saturday delivery.

8.2 Tumor cell purification and their chemosensitivity testing will be performed as per related DiaTech SOPs.

8.2.1 Tissue biopsy and effusion specimens will be treated to obtain a suspension containing single tumor cells and/or small cell aggregates composed of 2-20 tumor cells. Using gradient centrifugation, red blood cell lysing, cell strainers, magnetic beads and other appropriate techniques, the tumor cell suspension will be enriched to at least 80% purity and no less than 90% viability. Immunocytochemical stains or, when applicable, flow cytometry will be used to confirm the presence of specific tumor markers on purified cells After purification, selected chemotherapeutic agents will be tested against purified tumor cells in the MiCK assay.

8.2.2 The purified tumor cells will be suspended in culture medium and plated in 96-well microtiter plates. Multiple concentrations of chemotherapeutic agents will be achieved by adding each respective agent to wells in 5 μL aliquots The ranges of final drug concentrations will be based on reports of pharmacokinetic studies of the drugs and their active metabolites in patients. Data processing and quantification of drug-induced apoptosis will be performed by a proprietary ProApoTestTM software. The extent of apoptosis will be determined and expressed as kinetic units (KU) of apoptosis.

9.0 Efficacy measurement 9.1 For patients participating under Study Objective (2.1), the goal of the study is to establish a statistically significant discriminator of sensitivity which would correlate with the rate of CR. Such discriminator should be applicable to patient's populations participating under Study Objectives (2.1) and (2.2).

9.2 For patients participating under Study Objective (2.2), we would expect no greater than a 10% response rate in refractory solid tumor patients to any standard chemotherapy. A response rate to the MiCK assay-guided therapy of less than 10% would be of no further interest. A response rate of 10-30% will suggest the MICK assay needs further study. A response rate greater than 30% would justify usefulness of the MiCK assay in guiding chemotherapy of patients with refractory solid tumors.

10.0 Specimen's left over 10.1 If a specimen contains more tumor cells than needed for testing their sensitivity to the drugs specified by the patient's oncologist, an excess of the tumor cells may be considered for use for other research studies conducted by DiaTech Oncology. Patients will be asked for their permission to use specimen's left over for research purposes by signing the following release included in the requisition form: "You are participating in the Research Program which may result in improvements of the treatment outcome for cancer patients. There is no direct benefit for you at present time. Your physician is submitting to DiaTech a specimen containing your tumor cells. At DiaTech, we purify the tumor cells, count them, check their viability, and store them in the DiaTech Tissue Bank. All these procedures are performed at no cost to you or your family. Your cells may be used for the chemosensitivity testing for research purposes or in other studies. Results of the research may be published, or used commercially in the area of new anti-cancer drug or treatment protocol development. To assure your privacy, should the results of the studies be published, you will be referred to only by number. Your signature below indicates that you agree to these terms".

If a patient refuses to sign the above release, the specimen's left over will be decontaminated using 10% formaldehyde for 24h and discarded as per related SOP. If a patient grants his/her permission for use on the specimen's left over in a future research, an excess of the tumor cells will be frozen and stored in liquid nitrogen indefinitely.

10.2 Specimen's left over may be used to study anti-tumor effects of chemotherapeutic drugs or drug combinations, to study mechanisms of drug resistance, to correlate phenotypic features of the tumor cells with their drug sensitivity profile.

11.0 Plan of communication between Principal Investigator and co-Principal Investigator.

To insure proper communication between Vladimir Kravtsov, MD, the Study Principal Investigator, and participating co-Principal Investigator the following communication means will be used: FedEx delivery of the printed materials, Phone & Fax, E-mail, Video-conferencing

11.1 At the time of submission of the patient's specimen for the study, relevant clinical information will be submitted to DiaTech in the form of a study requisition form prepared by the participating co-PI (or designated staff nurse) using FedEx courier service.

11.2 Upon receiving the specimen and requisition form and after purification of tumor cells from the specimen, Dr. Kravtsov will place a telephone call to the referring oncologist (co-PI) to discuss the case.

11.3 Upon completion of the patient's tumor drug sensitivity testing, results will be scored and introduced to the study data base. Dr. Kravtsov will issue a study report and it will be faxed to the referring oncologist no later than 96h after receiving the specimen. After faxing the report, Dr. Kravtsov will call the referring oncologist to discuss the results.

11.4 After each 2 cycles of therapy, the patient's treatment response will be evaluated by the referring oncologists (co-PI). A study Response Evaluation Form (see attached) will be filled out and faxed to DiaTech to be included in the study data base.

11.5 After data from first ten consecutive patients are collected, a telephone or video conference will be scheduled between Dr. Kravtsov and the co-PI to summarize to discuss the preliminary results.

11.6 After data from first 30 consecutive patients are collected, an interim statistical analysis will be performed and Dr. Kravtsov will visit the participating hospital to present and discuss the results with the co-Principal investigator.

11.7 At the end of the first year, statistical analysis of the accumulated data will be performed and all participating co-PIs will be invited to a conference (place to be determined) to discuss the results.

11.8 DiaTech Study coordinator (Mr. Garry Latimer) will contact each site co-PI or a designated nurse monthly to assure proper supply of transportation containers and to address administrative issues.

11.9 All communication between the study coordinator and the participating oncology practice will be documented, reported to the Principal Investigator, and discussed with the co-Principal Investigator.

APPENDIX A

TREATMENT PLAN ALGORITHM FOR STUDY OBJECTIVE 2.1

Study Objective 2.1: To evaluate the ability of the MiCK assay to predict the outcome of chemotherapy of patients with solid tumors for first- and second-line treatments.

Chemotherapeutic agent(s) to be included in the treatment protocol are selected by a medical oncologist based on published standards and treatment guidelines.

Chemotherapy of the patient is initiated as per clinical treatment protocol and the oncologist discretion.

Name(s) of the drug(s) selected for the treatment is provided to the DiaTech lab along with the tumor material obtained from the patient.

Tumor cells purified from the patient's specimen are tested for their sensitivity to the drugs selected for the patient's treatment.

Results of the drug sensitivity testing are scored and introduced to the study database.

After each cycle of therapy, the patient is evaluated for the response to the treatment as per established criteria (clinical exam, CT, tumor markers).

Actual treatment response to the drug is compared with the drug scoring in the in vitro drug sensitivity test.

APPENDIX B

TREATMENT PLAN ALGORITHM FOR STUDY OBJECTIVE 2.2

Study objective 2.2: To evaluate the ability of the MiCK assay to guide chemotherapy of cancer patients in a third line, refractory treatment setting.

Chemotherapeutic agents available for the treatment are identified by a medical oncologist based on published standards and treatment guidelines.

Names of the drugs are provided to the DiaTech lab along with the tumor material obtained from the patient.

Tumor cells purified from the patient's specimen are tested for their sensitivity to the drugs selected by the patient's oncologist.

Results of the drug sensitivity testing are scored, introduced to the study database, and reported to the medical oncologist.

The drug with the best anti-tumor activity in the assay is used to treat the patient.

After each cycle of therapy, the patient is evaluated for the response to the treatment as per established criteria (clinical exam, CT, tumor markers).

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathological diagnoses of breast, lung, and ovarian adenocarcinomas and soft tissue sarcoma.
* Patients with de novo malignancies and no previous chemotherapy
* Patients with advanced refractory malignancies who received no more than 2 standard chemotherapy treatment protocols.
* Patients of any age group.
* Patients must have tumor which is accessible and agree to undergo biopsies, or drainage of effusions.
* Patients for whom chemotherapy is a treatment option.

Exclusion Criteria:

* Patients with symptomatic/uncontrolled parenchymal brain metastasis and non-accessible tumors.
* Patients with meningeal metastasis.
* Patients for whom chemotherapy is not clinically indicated.
* Pregnancy. During the course of the study, all patients of childbearing potential should be instructed to contact the treating physician if they suspect they might have conceived a child; for females, a missing or late menstrual period should be reported to the treating physician. If pregnancy is confirmed by a pregnancy test, the patient must not receive study medication and must not be enrolled into the study or, if already enrolled, must be withdrawn from the study. If a male patient is suspected of having fathered a child while on the study drugs, the pregnant female partner must be notified and counseled regarding the risk to the fetus. Pregnancy during the course of this study will be reported to the Principal Investigator as a serious adverse event. Women of childbearing potential are defined to include any female who has experienced menarche and has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not post-menopausal (defined as amenorrhea for more than 12 consecutive months); this also includes females using oral, implanted, or injectable contraceptive hormones, mechanical devices, or barrier methods to prevent pregnancy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-09; Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the ability of the MiCK assay to predict the outcome of chemotherapy of cancer patients | After chemotherapy
To evaluate the ability of the MiCK assay to guide chemotherapy of cancer patients | after chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Cary Presant, MD, Principal Investigator — Medical Director DiaTech Oncology; Pat Whitworth, MD, Principal Investigator — Director, Nashville Breast Center, PC; Alexander Zweibach, MD, PhD, Principal Investigator — Cancer Care Centers of South Texas; Karl Rogers, MD, Principal Investigator — Nashville Oncology Associates
Locations (3):
- United States (3):
  - Nashville Breast Center, Nashville, Tennessee
  - Nashville Oncology Associates, Nashville, Tennessee
  - Cancer Care Centers of South Texas, San Antonio, Texas